CLINICAL TRIAL: NCT06976996
Title: Efficacy of Subanesthetic Dose of Esketamine Combined With Different General Anesthetics on Quality of Early Postoperative Recovery in Patients Undergoing Painless Gastrointestinal Endoscopy
Brief Title: Efficacy of Esketamine Combined With Different General Anesthetics on Quality of Postoperative Recovery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Ju Gao, Study Director, Northern Jiangsu People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025ky074
Record Dates: First submitted 2025-05-02; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Quality of Postoperative Recovery
MeSH Terms: interventions — Saline Solution; Esketamine; Propofol; (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- group C (Placebo Comparator): normal saline (0.15 ml/kg) + ciprofol (0.5 mg/kg)
  Interventions: Drug: normal saline; Drug: ciprofol
- group E (Experimental): esketamine (0.15 mg/kg) + ciprofol (0.5 mg/kg)
  Interventions: Drug: esketamine; Drug: ciprofol
- group P (Experimental): esketamine (0.15 mg/kg) + propofol (2 mg/kg)
  Interventions: Drug: esketamine; Drug: propofol
- group EC (Experimental): esketamine (0.15 mg/kg) + etomidate-ciprofol (EC) mixture (0.2 ml/kg)
  Interventions: Drug: esketamine; Drug: etomidate-ciprofol (EC) mixture
- group EP (Experimental): esketamine (0.15 mg/kg) + etomidate-propofol (EC) mixture (0.2 ml/kg)
  Interventions: Drug: esketamine; Drug: etomidate-propofol (EP) mixture

INTERVENTIONS:
Drug: normal saline — normal saline (0.15 ml/kg)
  Arms: group C
Drug: esketamine — esketamine (0.15 mg/kg)
  Other Names: S-ketamine
  Arms: group E; group EC; group EP; group P
Drug: propofol — propofol (2 mg/kg)
  Arms: group P
Drug: etomidate-ciprofol (EC) mixture — etomidate-ciprofol (EC) mixture (0.2 ml/kg)
  Arms: group EC
Drug: ciprofol — ciprofol (0.5 mg/kg)
  Arms: group C; group E
Drug: etomidate-propofol (EP) mixture — etomidate-propofol (EP) mixture (0.2 ml/kg)
  Arms: group EP

SUMMARY:
To explore the effect of subanesthetic-dose esketamine combined with different general anesthetic drugs on the quality of postoperative recovery in patients undergoing painless gastrointestinal endoscopy.

DETAILED DESCRIPTION:
In this study, we planned to conduct a single-center, prospective, randomized, controlled, double-blind clinical trial to explore the effect of subanesthetic dose esketamine combined with different general anesthesia drugs on the postoperative recovery quality of patients undergoing painless gastrointestinal endoscopy combined with several commonly used intravenous general anesthesia drugs, aiming at gastroscopy combined with colonoscopy, a representative type of diagnosis and treatment of painless and comfortable anesthesia, and to provide more evidence-based medical evidence for clinical work.

ELIGIBILITY:
Inclusion Criteria:

* (1) Aged between 18 and 75 years old (inclusive); (2) ASA (American Society of Anesthesiologists) physical status classification of Class I to III; (3) Body Mass Index (BMI) ranging from 18 to 30 kg/m²; (4) Individuals scheduled to undergo combined gastroscopy and colonoscopy under painless anesthesia; (5) Those with a patent airway and no history of difficult intubation or difficult airway management; (6) Individuals with intact cognitive function, who have provided informed consent, voluntarily participate in this study, and are capable of cooperating to complete data collection.

Exclusion Criteria:

* （1）A history of unregulated diabetes mellitus, hypertension, or hypotension; （2）Concomitant hyperthyroidism or hypothyroidism; （3）Concomitant psychiatric or neurological disorders; （4）Severe hepatic or renal insufficiency; （5）Concomitant glaucoma, severe hearing or visual impairment that hinders cooperation; （6）Individuals with significant organ dysfunction; （7）Those with allergies to or contraindications for the study drug; （8）Patients with aneurysmal vascular diseases involving the thoracic or abdominal aorta, intracranial arteries, or peripheral arterial vessels; （9）Individuals who are unable to cooperate in completing the Quality of Recovery-15 (QoR-15) questionnaire.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-03-16 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery-15 | Postoperative day 1 and 3
  The QoR-15 (Quality of Recovery-15) evaluates the quality of recovery across five dimensions: physical comfort (50 points), emotional state (40 points), physical independence (20 points), psychological support (20 points), and pain (20 points). The total score of the QoR-15 ranges from 0 (indicating the poorest quality of recovery) to 150 (representing the best quality of recovery).

SECONDARY OUTCOMES:
Perioperative vital signs | Perioperative
  The following parameters: Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP), Mean Arterial Pressure (MAP), Heart Rate (HR), and Peripheral Oxygen Saturation (SpO₂) were measured and recorded at the following time points: before anesthesia induction (T0), immediately after anesthesia induction (T1), at the moment when the gastroscope entered the larynx (T2), when the gastroscope was withdrawn from the pharyngeal cavity (T3), when the colonoscope entered the anus (T4), and at the completion of colonoscopy (T5).
Anesthesia Recovery Time | during surgery and arrived at PACU (up to 30 minutes after surgery)
  The time interval between the last administration of general anesthetic agent(s) and the moment when the patient achieves a Modified Aldrete Score of ≥9.
Procedure Duration | during surgery and arrived at PACU (up to 30 minutes after surgery)
  From the beginning of gastroscopy to the end of colonoscopy withdrawal
PACU residence time | during surgery and arrived at PACU (up to 30 minutes after surgery)
  The time from entering the PACU to leaving the PACU after the end of gastroscopy combined with colonoscopy;
Anesthetic drug use | during surgery and arrived at PACU (up to 30 minutes after surgery)
  Total amount of sedative medication used, number of cases of norepinephrine, and number of cases of remifentanil.
The way the patient leaves the endoscopy center | Postoperative
  The way in which the patient is discharged from the PACU after the anesthesia resuscitation is up to standard;
The length of the patient's stay in the hospital after leaving the endoscopy center in the PACU | Postoperative
  The length of the patient's stay in the hospital from the time the patient leaves the PACU until he leaves the hospital.
The way the patient leaves the hospital | Postoperative
  The patient's method of leaving the hospital, such as walking on their own, driving any means of transportation, etc.
Satisfaction score | Postoperative
  Patient, anesthesiologist, and digestive endoscopist satisfaction with the whole gastroscopy combined with colonoscopy. Using the NRS, eleven numbers from 0-10 represent satisfaction, with 0 being dissatisfied and 10 being the most satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Jiangsu People's Hospital, Yangzhou, Jiangsu, China